CLINICAL TRIAL: NCT02031835
Title: Body Weight Supported Treadmill Training as Physical Therapy Treatment to Spinal Cord Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Avraam Ploumis, Principal Invastigator, University of Ioannina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UIoannina612014
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Spinal Cord Injury/Damage
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BWSTT (3 days a week for maximum of 20 minutes session) (Other): BWSTT (20 minutes of treadmill training (velocity (≥0.1km/h) and body weight support (≤40% of patients weight) according to patients capability and comfort
  Interventions: Procedure: BWSTT (3 days a week for maximum of 20 minutes session)

INTERVENTIONS:
Procedure: BWSTT (3 days a week for maximum of 20 minutes session)

SUMMARY:
The purpose of this current prospective study is to assess the effects of body weight support treadmill training (BWSTT) in individuals with spinal cord injury (SCI). Training intervention aim at improving: quality of life, walking capability, spasticity, functions in every day life, bone mass density and related hematological factors. The examination consisted of (1) neurological classification by ASIA standard neurological classification of spinal cord injury working sheet, (2) spasticity evaluation of lower limbs by Modified Ashworth Scale, (3) walking independence evaluation by Walking Index for Spinal Cord Injury II (WISCI II), (4) patient's quality of life perspective by World Health Quality of Life- BREF (WHOQOL-BREF), (5) the functional status by 10-item Modified Barthel Index, (6) bone mass density (BMD) by Dual-energy X-ray absorptiometry (DXA) scan, (7) body tissue consistency by full body DXA scan, (8) skeletal system health associated blood factors (calcitonin, osteocalcin, 25 OH vitamin D, 1,25- (OH)2 vitamin D, ostase and parathyroid hormone) by hematological tests. The results will be collected and evaluated using statistical software (i.e. SPSS).

ELIGIBILITY:
Inclusion Criteria:

* SCI
* ASIA classification B, C or D
* clinical stable

Exclusion Criteria:

* unstable cardiac conditions
* epilepsy
* autonomic dysreflexia
* significant musculoskeletal problems in lower extremities other than SCI
* Parkinson's disease

Ages: 8 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2012-03; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
WISCI II | At the time of Admittance to the rehabilitation department (at baseline) and after six weeks
  Change of walking independence at six weeks

SECONDARY OUTCOMES:
ASIA standard neurological classification for spinal cord injury patients working sheet | At the time of Admittance to the rehabilitation department (at baseline) and after six weeks
  Change of neurological impairment status at six weeks
Modified Ashworth scale | At the time of Admittance to the rehabilitation department (at baseline) and after six weeks
  Change of spasticity of leg muscles at six weeks
WHOQOL-BREF | At the time of Admittance to the rehabilitation department (at baseline) and after six weeks
  Change of patients' perspective of life quality at six weeks
10-item Modified Barthel Index | At the time of Admittance to the rehabilitation department (at baseline) and after six weeks
  Change of function at six weeks
DXA scan | At the time of Admittance to the rehabilitation department (at baseline) and after six weeks
  Change of BMD of hip and spine at six weeks
Full Body DXA scan | At the time of Admittance to the rehabilitation department (at baseline) and after six weeks
  Change of body tissue consistency at six weeks
Hematological analysis | At the time of Admittance to the rehabilitation department (at baseline) and after six weeks
  Change of blood's calcitonin, osteocalcin, 25 OH vitamin D, 1,25- (OH)2 vitamin D, ostase and parathyroid hormone concentrations at six weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece